CLINICAL TRIAL: NCT06794983
Title: Health Systems Innovations for Supporting Transitions of Care for Incarcerated People Living With Substance Use Disorders
Brief Title: Calls and Coordination for Transitions of Care at Re-entry
Acronym: Call2Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1669; 2R01DA047889-06 (NIH); A538500 (Other: UW Madison); Protocol Version 11/8/2024 (Other: UW Madison); SMPH/POP HEALTH SCI/POP HLTH (Other: UW Madison)
Record Dates: First submitted 2025-01-23; First posted 2025-01-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Prisoners; Substance Use History; Chronic Medical Conditions; Psychiatric Condition; Substance Use Disorder (SUD)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Group (Experimental): Participants will receive phone calls and texts.
  Interventions: Other: In-person visit with study team member; Other: Phone calls and texts
- Phone + Nurse Case Manager (NCM) Group (Experimental): Participants will work with a nurse case manager, who will call and text.
  Interventions: Other: In-person visit with NCM; Other: Phone calls and texts - NCM

INTERVENTIONS:
Other: In-person visit with study team member — Participants meet with a study team member before they are released from prison.
  Arms: Phone Group
Other: In-person visit with NCM — Participants meet with a NCM before they are released from prison.
  Arms: Phone + Nurse Case Manager (NCM) Group
Other: Phone calls and texts — Study team member calls and texts participants after they are released from prison.
  Arms: Phone Group
Other: Phone calls and texts - NCM — Nurse case manager calls and texts participants after they are released from prison.
  Arms: Phone + Nurse Case Manager (NCM) Group

SUMMARY:
The goal of this clinical trial is to learn if a short program for people being released from prison can help connect them to medical care. The main question it aims to answer is:

* Will there be more non-emergency, outpatient clinic visits?

Researchers will compare the number of clinic visits between people who use a Nurse Case Manager (NCM) to people in enhanced usual care.

Participants will:

* Complete surveys
* Talk to a study team member 2-3 times, or talk to a study team member 2-3 times and talk to an NCM 6-11 times

DETAILED DESCRIPTION:
The objective of this clinical trial is to test the effectiveness of a transitional care program adapted to meet the healthcare needs of adults after release from prison. The goal of the transitional care intervention being tested is to help the study participants connect to primary care within 60 days of release through weekly check-in calls. Participants in this study are enrolled approximately 6 months before their anticipated release. One group will receive weekly phone calls for up to 60 days post-release. Additionally, novel, linked administrative datasets will be leveraged to enhance, contextualize, and clarify policy implications of the clinical trial results.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* eligibility for WI Medicaid and intention to enroll before release
* substance use history (i.e., "have you ever considered your alcohol or drug use to be a problem?"), and
* living with, or history of, a chronic medical or psychiatric condition other than substance use disorder. This is defined as ever having been diagnosed with a medical or psychiatric chronic condition, or currently taking prescription medications for a chronic condition.
* able to read, understand, and speak English.

Exclusion Criteria:

* ineligible for WI Medicaid
* no substance use history
* not living with, or no history of, chronic medical or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who attend a Non-Emergency Outpatient Visit within 60 Days of Release From Prison | 2 months post-release, approximately 5 months on study

SECONDARY OUTCOMES:
Number of participants who attend a Non-Emergency Outpatient Visit for Substance Use Disorder within 60 Days of Release From Prison | 2 months post-release, approximately 5 months on study

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite Burns, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes